CLINICAL TRIAL: NCT00387907
Title: Open Label, Uncontrolled, Study of XRP9881 (Larotaxel) in Combination With Weekly Trastuzumab (Herceptin®) in Patients With HER2 Positive Metastatic Breast Cancer (MBC)
Brief Title: Study of Larotaxel in Combination With Weekly Herceptin® in Patients With HER2 Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD10037; XRP9881
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Advanced Breast Cancer; Breast Cancer; Metastatic Breast Cancer
Keywords: Herceptin; Taxane; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — larotaxel; Trastuzumab

ARMS (1):
- Larotaxel + Trastuzumab (Experimental)
  Interventions: Drug: larotaxel (XRP9881); Drug: trastuzumab

INTERVENTIONS:
Drug: larotaxel (XRP9881) — administered as a 1-hour IV infusion on Day 1 of every 3 weeks (q3w)
Drug: trastuzumab — administered as a 90-minute IV infusion on Day 1 of every week (qw)

SUMMARY:
The purpose of this study is to evaluate the anti-tumor activity of the combination of experimental drug (larotaxel) when combined with Herceptin® in patients with advanced breast cancer. Anti-tumor activity will be determined by looking at changes in tumor size on CT or MRI scans. Additional goals of this study are to look at patient safety, to determine how long the study drugs (larotaxel and Herceptin®) stay in the patient's body and what effects the study medications may have on each other, and to find out how long patients remain cancer free on this study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer
* Evidence that cancer has spread beyond its original location or has come back and cannot be removed by surgery
* No more than one prior treatment for advanced disease
* Her2 positive status
* Adequate liver and kidney function
* No remaining severe harmful effects to prior treatments

Exclusion Criteria:

* Certain heart condition
* Pregnant Women
* History of another cancer except some skin cancers and cervical cancer
* Taking other treatments for your cancer at the time you enter the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Tumor response measured | every 2 cycles during treatment phase

SECONDARY OUTCOMES:
Progression Free Survival and Overall Survival | measured every 3 weeks during study treatment, then every 6 weeks after a patient has stopped the study treatment until the patient's cancer worsens, then every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Winer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Sanofi-Aventis Administrative Office, Malvern, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com